CLINICAL TRIAL: NCT06707493
Title: A Randomized, Placebo-Controlled Phase 2 Study of IDH1 Inhibition Using Ivosidenib as Maintenance Therapy for IDH1-mutant Acute Myeloid Leukemia Following Allogeneic Stem Cell Transplantation
Brief Title: Ivosidenib as Post-HSCT Maintenance for AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Amir Fathi, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-641
Record Dates: First submitted 2024-11-23; First posted 2024-11-27 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: IDH1 Mutation; Acute Myeloid Leukemia (AML); Hematopoietic Stem Cell Transplant (HSCT)
Keywords: hematopoietic stem cell transplantation (HCT); IDH1-mutant acute myeloid leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ivosidenib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivosidenib (Experimental): After screening and standard of care hematopoietic stem cell transplantation (HCT) and any standard treatment before and after the HSCT, Ivosidenib will be given orally (PO) once daily (QD) in 28-day continuous cycles. Ivosidenib is administered at a pre-determined dose with a goal of 500mg daily. Participants begin study treatment 45 to 90 days after HCT, and treatment will continue for up to 24 months. Study visits and assessments occur throughout study treatment and in follow-up. After the 24-month treatment period, participants are followed for up to 12 additional months.
  Interventions: Drug: Ivosidenib
- Placebo (Placebo Comparator): After screening and standard of care hematopoietic stem cell transplantation (HCT) and any standard treatment before and after the HSCT, Placebo will be given orally (PO) once daily (QD) in 28-day continuous cycles. Participants begin study treatment (placebo) 45 to 90 days after HCT, and treatment (placebo) will continue for up to 24 months. Study visits and assessments occur throughout study treatment period and in follow-up. After the 24-month treatment period, participants are followed for up to 12 additional months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivosidenib — Ivosidenib tablets are supplied as 50 mg, 200 mg, and 250 mg strengths, to be taken orally.
  Other Names: AG-120; S95031
  Arms: Ivosidenib
Drug: Placebo — Placebo tablets are taken orally.
  Arms: Placebo

SUMMARY:
This is a Phase 2 study of the study drug, ivosidenib (a mutant IDH1 inhibitor), compared to placebo, given to patients with IDH1-mutant acute myeloid leukemia (AML) after hematopoietic stem cell transplantation (HCT).

DETAILED DESCRIPTION:
This is a prospective, placebo-controlled, randomized, single-blinded, multi-center, phase II study of the mutant IDH1 inhibitor, ivosidenib, compared to placebo in participants with AML after HCT. This study is examining whether or not ivosidenib is beneficial as an agent to prevent the relapse of IDH1-mutated acute myeloid leukemia after hematopoietic stem cell transplantation. The U.S. Food and Drug Administration (FDA) has not approved ivosidenib for this indication following HCT but it has been approved for other uses.

The research study procedures include screening for eligibility and study treatment including evaluations and follow-up. The HCT and any standard treatment before and after the HCT is standard of care.

The estimated length of participation in the study is 3.5 years from screening to the end of planned follow-up, including up to 24 months of study treatment. After the 24-month period, participants are followed for up to 12 additional months. It is expected that about 75 people will take part in this research study.

Servier, a pharmaceutical company, is supporting this research study by providing ivosidenib/placebo and funding for research activities.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of IDH1(R132)-mutant acute myeloid leukemia (AML). IDH1 mutations could have been detected by any mutational technique at any prior point including at diagnosis or remission.
* Between the ages of 18 and 75 years
* Will undergo allogeneic hematopoietic stem cell transplantation (HSCT) for their malignancy. Conditioning may be either conventional myeloablative (MAC) or reduced intensity conditioning (RIC). There will be no restrictions on type of graft source.
* ECOG performance status ≤ 2
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1000/µL without growth factor support (e.g. GCSF) in the previous 7 days.
  * Platelet count ≥ 50,000/µL without transfusional support in the previous 7 days.
  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 3x institutional upper limit of normal (ULN)
  * Direct bilirubin < 2.0 mg/dL
  * Calculated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula)
* LVEF must be equal to or greater than 40%, as measured by MUGA scan or echocardiogram
* Female patients of childbearing potential must have a negative pregnancy test
* The effects of ivosidenib on the developing human fetus are unknown. For this reason female participants of child-bearing potential and male participants must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during the entire study treatment period and through 90 days after the last dose of treatment
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplants.
* Morphologically relapsed or refractory disease, as assessed by bone marrow aspirate and biopsy performed within 42 days prior to study entry
* History of other malignancy(ies) unless

  * the participant has been disease-free for at least 5 years and is deemed by the investigator to be at low risk of recurrence of that malignancy, or
  * the only prior malignancy was cervical cancer in situ and/or basal cell or squamous cell carcinoma of the skin
* Known diagnosis of active hepatitis B or hepatitis C
* Current or history of congestive heart failure New York Heart Association (NHYA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF < 40%, as measured by MUGA scan or echocardiogram)
* Current or history of ventricular or life-threatening arrhythmias or diagnosis of long-QT syndrome
* QTc interval (i.e., Friderica's correction [QTcF]) ≥ 450 ms or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening
* Uncontrolled intercurrent illness that would limit compliance with study requirements.

Post-transplantation Pre-Treatment Criteria Treatment may begin at any time between day 45 and day 90 following stem cell transplantation.

However, at time of treatment start, it must be ensured that:

* The patient has continued willingness and interest in participating in the study.
* There is no systemic infection requiring IV antibiotic therapy within 7 days preceding the first dose of study drug, or other severe infection
* Chimerism studies reveal that ≥ 70% of blood or bone marrow cells, or of the CD33 expressing fraction, are of donor origin,
* There is no acute graft versus host disease (GVHD), requiring an equivalent dose of ≥ 0.5mg/kg/day of prednisone within one week of starting ivosidenib / placebo, or have escalation of systemic immunosuppression in terms of increase of corticosteroids or addition of new agent/modality within two weeks of starting ivosidenib / placebo.
* For prophylaxis for GVHD, agents that are permitted for administration on study:

  * Tacrolimus
  * Cyclosporine
  * Sirolimus
  * Cyclophosphamide
  * Mycophenolate Mofetil
  * Methotrexate
  * ATG
  * Ruxolitinib
  * Vedolizumab
  * As standards of care may change, any other prophylactic agents used should be discussed with the PI.
* Investigational agents, defined as not approved for any indication, are forbidden unless the participant comes off study.

  * Agents used to treat GVHD that are permitted for administration on study:
  * Any agent used in prophylaxis may be continued (see list above)

    * Ruxolitinib
    * Etanarcept
    * ATG
    * Belumosidil
    * Axatilimab
    * Rituximab
    * Fecal microbiota transplantation
    * Alpha1-Antitrypsin
    * Pregnyl
    * Extracorporal photopheresis (ECP)
  * As standards of care may change, any other treatment agents used should be discussed with the PI.
  * Investigational agents, defined as not approved for any indication, are forbidden unless the participant comes off study.
* There is no evidence of relapsed/recurrent/residual disease.
* Prior to the start of ivosidenib / placebo administration, the participant must have adequate hematological function, defined as:

  * ANC ≥ 1000/µL
  * Platelets ≥ 50,000/µL

and adequate organ function defined as

* Direct bilirubin level < 2.0 mg/dL
* AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 3x institutional upper limit of normal (ULN)
* No presence of congestive heart failure, defined by New York Heart Association (NHYA) criteria as class 3 or 4
* Calculated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival (RFS) | Time of randomization to 24 months post-randomization, death, or disease relapse whichever occurs first.
  Relapse-Free Survival is defined as the time from randomization following transplant to disease relapse or death due to any cause, whichever occurs first. Participants alive without relapse are censored at the date of last seen alive. The primary analysis will be performed using the Kaplan-Meier method with log-rank test.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 39 months (Day of HCT (Day -90 to Day -45) through 24 months of treatment period and 12 months of follow-up)
  Overall Survival is defined as the time from stem cell transplant (HCT) to the date of death due to any cause. Participants who are alive at the analysis / cutoff date will be censored at the last contact date. Baseline characteristics will be reported descriptively and compared using Fisher's exact test, χ2 test or Wilcoxon rank-sum test, as appropriate. The Kaplan-Meier method will be used to estimate OS; Multivariable Cox regression analysis will be used for OS analysis.
Incidence of treatment related adverse events (TRAE) | Up to 25 months (Day 1 of study drug treatment for up to 24 months of treatment plus 30 days post final dose)
  TRAEs will be graded and categorized using the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5. Baseline characteristics will be reported descriptively and compared using Fisher's exact test, χ2 test or Wilcoxon rank-sum test, as appropriate.
Cumulative incidence of acute and chronic Graft vs. Host Disease (GVHD) | Up to 36 months (Start of study treatment for 24 months, plus 12 months of follow-up)
  Chronic GVHD will be assessed as per the National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease. Cumulative incidence of acute and chronic GVHD (grade II-IV acute GVHD, grade III-IV acute GVHD, chronic GVHD, steroid-requiring chronic GVHD) will be estimated in the context of a competing risks framework. Gray test and Gray regression analysis will be used for comparison of cumulative incidence of GVHD.
Measurable Residual Risease (MRD) | Pre-transplant screening (up to Day -132) through 12 months of study treatment period, for up to 16.5 months.
  MRD will be assessed by Next Generation Sequencing (NGS) testing at screening before stem cell transplant, post-transplant before initiation of study treatment, and at the start of study treatment cycles 6 and 12.
Cumulative incidence rate of relapse of acute myeloid leukemia (AML) | From stem cell transplant through 12 months treatment period or relapse, whichever is first., up to 15 months.
  Disease assessment (relapse) will be based on modified IWG criteria or other appropriate response criteria for the malignancy being studied. Cumulative incidence of relapse of AML will be estimated in the context of a competing risks framework using the Gray test and Fine and Gray regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Amir T Fathi, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [Amir T. Fathi, M.D. afathi@mgh.harvard.edu ]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation